CLINICAL TRIAL: NCT04484701
Title: 68Ga-PSMA-11 Positron Emission Tomography / Computed Tomography (PET/CT) for Assessment of High Risk or Recurrent Prostate Cancer
Brief Title: [68Ga]Ga-PSMA-11 PET/CT in the Assessment of High Risk and Recurrent Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H20-01325
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasm; Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PSMA-11 PET/CT scan: All participants will undergo the same procedures listed in "Detailed Description" in the protocol section.
  Interventions: Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — PET/CT scan with radiotracer 68Ga-PSMA-11

SUMMARY:
Prostate cancer is the third most common cause of cancer death in men. Most patients with localized prostate cancer will be cured with surgery or radiation therapy, but up to 35% of patients will have their prostate cancer return. Whether it has returned locally or distantly determines which type of treatment they will receive. Current conventional imaging modalities have limitations particularly at low prostate specific antigen levels. This study proposes to use Gallium-68-PSMA-11 (68Ga-PSMA-11) Positron Emission Tomography / Computer Tomography (PET/CT) scans which targets prostate-specific membrane antigens (PSMA) to detect where in the body the prostate cancer has recurred.

DETAILED DESCRIPTION:
This is a prospective registry study to evaluate the diagnostic utility of 68Ga-PSMA-11 PET/CT to stage patients with high risk prostate cancer, localize sites of biochemical recurrence of prostate cancer, and restage patients with advanced prostate cancer before and after onset of new therapy.

Eligible subjects will undergo a 68Ga-PSMA-11 PET/CT at the British Columbia Cancer (BCC) - Vancouver. Each subject will receive a 68Ga-PSMA-11 PET/CT scan at the BCC - Vancouver, as part of this research study. Each study subject will receive a bolus intravenous dose of 68Ga-PSMA-11. The subject will rest in a comfortable chair for 60 minutes and will then be taken to the PET/CT scanner for images. The PET/CT scan will take approximately 2.5 hours of patient time above and beyond the time needed for standard of care.

Medical History Questionnaire: Demographic and medical history data will be collected either in person before the PET scan appointment or by mail or phone, whichever is the most convenient to the subject.

Follow-up assessments: All subjects will be contacted by phone the day after the injection of 68Ga-PSMA-11. The subjects will be asked if they experienced any undesirable effects during the 12 hours after the administration of 68Ga-PSMA-11. The local site attending nuclear medicine physician will then make an assessment as to whether these effects are likely related to 68Ga-PSMA-11 administration.

All subjects will be followed for 5 years following the 68Ga-PSMA-11 PET/CT exam to assess the presence of recurrence. The evaluation will include a chart review of available imaging, laboratory tests, and treatment. The data required can be obtained from a review of the patient's paper and electronic charts, supplemented by telephone contact as needed to complete the information.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 2 or less.
* Subjects with high risk prostate cancer (CAPRA score 6 or higher) being considered for curative-intent surgery or radiation therapy (including brachytherapy)
* Subjects with biopsy confirmed prostate cancer being considered for curative-intent surgery or radiation therapy (including brachytherapy), who have unconfirmed suspicious findings on conventional medical imaging staging examinations.
* Subjects with biochemical recurrence or persistence of prostate cancer following initial curative treatment by radical prostatectomy, with two consecutive PSA values >0.2 ng/ml measured more than 6 weeks after radical prostatectomy. If subjects received subsequent systemic therapy, the most recent PSA measurement prior to PET/CT imaging must be greater than 0.2 ng/mL.
* Subjects with biochemical recurrence or persistence of prostate cancer following initial curative treatment by radical prostatectomy and subsequently treated by salvage radiotherapy or pelvic node dissection, with two consecutive PSA values >0.2 ng/ml. If subjects received subsequent systemic therapy, the most recent PSA measurement prior to PET/CT imaging must be greater than 0.2 ng/mL.
* Subjects with biochemical recurrence of prostate cancer after initial curative therapy with radiation therapy (including brachytherapy), or non-standard local ablative therapy (such as high frequency ultrasound, cryoablation, focal laser ablation, etc.), with a PSA level >2 ng/mL above the nadir after radiation therapy.
* Subjects with advanced castration sensitive or castration resistant prostate cancer being considered for localized treatment (surgery, brachytherapy, radiotherapy) of recurrent or oligometastatic prostate cancer. Castration resistance is defined as a PSA level > 1.0 ng/mL, with 2 consecutive rises above the nadir, in the presence of castrate levels of testosterone (< 1.7 nmol/L).
* Subjects with metastatic or castration resistant prostate cancer being evaluated for systemic therapy administered in therapeutic clinical trials. The PSA level must be > 1.0 ng/mL, with 2 consecutive rises above the nadir, in the presence of castrate levels of testosterone (< 1.7 nmol/L).

Exclusion Criteria:

* Medically unstable (e.g. acute illness, unstable vital signs)
* Unable to lie supine for the duration of imaging
* Unable to provide written consent
* Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)

Exclusion criteria for the use of furosemide Subjects can still participate in the research study and undergo the [68Ga]Ga-PSMA-11 scan if they are unable or unwilling to receive a furosemide injection.

* Subjects with end stage renal disease.
* Subjects with documented history of severe progressive chronic kidney disease (glomerular filtration rate less than 30 mL/min/1.73 m2).
* Subjects with hypersensitivity to furosemide (Lasix).
* While cross-reactivity between sulfonamide antibiotics and non-antibiotics has been disproven, subjects who have a history of sulfonamide antibiotics or sulfonylureas may be at a higher risk of allergic reaction to furosemide due to a higher general predisposition to allergic reactions. In those instances, the administration of furosemide is left at the discretion of the local site investigator after discussion with the study subject.
* Subjects with severe hypokalemia, hyponatremia, hypovolemia, dehydration or hypotension.
* Subjects with untreated bladder outlet obstruction or lower urinary tract symptoms, who have a history of obstructive episodes that required hospitalization, emergency department visits and/or bladder catheterization for relief of symptoms.

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with high risk prostate cancer at initial presentation (CAPRA score 6 or higher), subjects with biochemical persistence of prostate cancer following radical prostatectomy, subjects with biochemical recurrence of prostate cancer following initial curative treatment with radical prostatectomy or radiation therapy, subjects with biochemical recurrence of prostate cancer following radical prostatectomy who received subsequent salvage radiotherapy, and subjects with advanced prostate cancer (castration sensitive or castration resistant disease that is metastatic with conventional imaging, castration resistant disease that is non-metastatic on conventional imaging).
Sampling Method: Non-Probability Sample
Enrollment: 1574 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-PSMA-11 PET/CT imaging in the assessment of high risk and recurrent prostate cancer. | 5 years after PSMA-11 PET/CT scan
  Determination of sensitivity when compared with pathology reports (if available) and routine imaging (CT, MRI, bone scan) if available.

SECONDARY OUTCOMES:
Predictive value of 68Ga-PSMA-11 PET/CT imaging | 5 years after the PSMA PET scan
  The clinical predictive value will be assessed by multivariate analysis, using a Cox proportional hazard model, including established clinical parameters at initial presentation or relapse for the 5 most active lesions.
Accuracy of 68Ga-PSMA-11 PET/CT imaging | 5 years after the PSMA PET scan
  The accuracy (along with the confidence interval) of 68Ga-PSMA-11 will be calculated for subjects with an available gold standard.
  The gold standard for the detection of lesions will be established through a combination of: 1) pathology results following surgical resection; 2) disease progression of specific 68Ga-PSMA-11 findings on clinical or conventional imaging follow-up; 3) unequivocal disease response of specific 68Ga-PSMA-11 findings on conventional imaging follow-up after treatment; 4) decrease of PSA level after targeted radiation of 68Ga-PSMA-11 findings; 5) progression of 68Ga-PSMA-11 findings on subsequent 68Ga-PSMA-11 imaging associated with a concurrent increase in PSA level; 6) regression of [68Ga]Ga-PSMA-11 findings on subsequent [68Ga]Ga-PSMA-11 imaging associated with a concurrent decrease in PSA level.
Specificity of 68Ga-PSMA-11 PET/CT imaging | 5 years after the PSMA PET scan
  The specificity (along with the confidence interval) of [68Ga]Ga-PSMA-11 will be calculated for subjects with an available gold standard (see above for definition).
Number of participants with self-reported 68Ga-PSMA-11-related adverse event | 12 hours post 68Ga-PSMA-11 injection
  Patients will be contacted by phone the day after the 68Ga-PSMA-11 PET/CT scan to see if they experienced any adverse events in the 12 hours following the 68Ga-PSMA-11 injection. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No plan.